CLINICAL TRIAL: NCT03007862
Title: Salivary Alpha Amylase Bronchial Measure for Early Aspiration Pneumonia Diagnosis in Patients Treated With Therapeutic Hypothermia After Out-of-hospital Cardiac Arrest.
Brief Title: Bronchial Alpha Amylase as a Marker for Early Aspiration Pneumonia in Therapeutic Hypothermia.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-37
Record Dates: First submitted 2016-12-28; First posted 2017-01-02 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2016-12

CONDITIONS: Early Aspiration Pneumonia
MeSH Terms: conditions — Pneumonia, Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Early Aspiration Pneumonia is a frequent and dreadful complication in survivors of cardiac arrest. Therapeutic Hypothermia widely used in Intensive Care Unit for its benefice on post cardiac arrest syndrome may otherwise hide signs of early pneumonia that may occur without use of a reliable screening biological marker. The goal is to assess the diagnostic accuracy of bronchial alpha amylase measure to predict a risk of early aspiration pneumonia in patients successfully resuscitated after out-of-hospital cardiac arrest.

In this prospective non interventional study we included patients resuscitated after cardiac arrest and treated with Targeted Temperature Management (TTM). A distal bronchoalveolar lavage using specific display (Combi-Cath) was executed immediately after admission for each patient with both biochemic and bacteriological analysis including dosage of bronchial salivary alpha amylase. Urea was used as a marker of dilution in the measure of bronchial and plasmatic alpha amylase. Aspiration pneumonia diagnosis was established with clinical and biological criteria. On this basis we intended to determine a threshold measure of alpha amylase predicting occurrence of aspiration pneumonia and allowing a guidance in antibiotherapy prescription. Sensibility and Specificity of this technique were determined.

ELIGIBILITY:
Inclusion Criteria:

* Well resuscitated patients after out-of-hospital cardiac arrest
* Indication of Therapeutic Temperature Management
* Patients aged over 18 years
* Immediate or deferred acceptation of study

Exclusion Criteria:

* Patients aged under 18 years.
* Pregnant women.
* Against indication to therapeutic hypothermia.
* Active therapeutic limitation after admission.
* Patient without social security.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early Aspiration Pneumonia after out-of-hospital cardiac arrest treated with Therapeutic Temperature Management
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Early Aspiration Pneumonia | Within 5 days
  Diagnosis of aspiration pneumonia after cardiac arrest with clinical, biological and radiological criteria including fever, leucocytes, broncho alveolar secretion, chest radiography and bacteriological identification.

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France